CLINICAL TRIAL: NCT06550622
Title: Improved Sensitivity Detection of Serum HBsAg in Chronic Hepatitis B Patients Achieving Functional Cure and Its Association With HBsAg Reversion
Brief Title: Improved Sensitivity Detection of Serum HBsAg and HBsAg Reversion
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, Professor, Huashan Hospital
Other Study IDs: 2024-700
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis B, Chronic
Keywords: HBsAg next assay; Functional cure; HBsAg loss; HBsAg reversion
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: CHB patients with HBsAg level<0.005 IU/mL
- Group B: CHB patients with 0.005 IU/mL< HBsAg level < 0.05 IU/mL

SUMMARY:
The goal of this observational study is to learn about the HBsAg reversion rate at 48 weeks off treatment in HBsAg-negative patients by HBsAg NEXT assay which has improved sensitivity compared to current ARCHITECT HBsAg Assay.

The main question it aims to answer is:

What's the HBsAg reversion rate at 48 weeks off treatment in HBsAg-negative patients by HBsAg NEXT assay? HBsAg NEXT assay technology (lower limit of detection for HBsAg is 0.005 IU/ml) and current ARCHITECT HBsAg assay (lower limit of detection for HBsAg is 0.05 IU/ml) are applied for HBsAg detection in patients achieving functional cure, and to compare the difference in HBsAg reversion rate 48 weeks off treatment under the two types of criteria.

DETAILED DESCRIPTION:
In this study, chronic hepatitis B patients who achieved HBsAg loss by current ARCHITECT HBsAg testing (lower limit of detection for HBsAg is 0.05 IU/ml) under interferon therapy and received consolidation therapy for 3 month after that were screened for eligibility. Those who are willing to discontinue were enrolled in the study. Patients were divided in two groups according to HBsAg levels，one with patients who were HBsAg-negative （HBsAg<0.005 IU/mL）by HBsAg next assay , and the other with patients who had HBsAg levels between 0.005 IU/mL and 0.05IU/mL. Patients were followed up for 48 weeks after discontinuation after HBsAg loss and HBsAg reversion rates in the two groups were analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-negative by Abbott's HBsAg Test and HBeAg-negative;
* Having serum specimens retained at baseline and at 48 weeks off treatment follow up;
* Being willing to follow up regularly for 1 year.

Exclusion Criteria:

* Patients with hepatitis B cirrhosis in the compensated and decompensated stages: this includes patients with a clear history of cirrhosis (imaging or histological evidence) or Child-Pugh score ≥5 prior to NUC treatment, or who have had complications of the decompensated stage of cirrhosis, such as ascites, hepatic encephalopathy, or ruptured oesophago-gastric fundal varices bleeding;
* Combined HAV, HCV, HDV, HEV, HIV infections, alcoholic liver disease, inherited metabolic liver disease, pharmacological liver disease, non-alcoholic fatty liver disease, autoimmune liver disease and other chronic liver diseases;
* Primary hepatocellular carcinoma or those with AFP greater than 100 ng/ml at screening and imaging suggestive of possible malignant hepatic occupancy; or patients with AFP greater than 100 ng/ml for a sustained period of 3 months;
* Patients with a combination of other malignant tumours (excluding those who have been cured);
* Patients with severe diseases or uncontrolled disease
* Those who are also participating in other clinical studies;
* Patients deemed unsuitable by the investigator to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject studied were HBsAg-negative, HBeAg-negative, and anti-HBe positive patients with chronic hepatitis B
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2027-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
HBsAg reversion rate | 48 weeks
  HBsAg reversion rate in patients with HBsAg loss by Abbott's HBsAg next assay at week 48 off treatment

SECONDARY OUTCOMES:
Proportion of patients who were HBsAg positive | 48 weeks
  Proportion of patients who were HBsAg positive by HBsAg Next assay in those who were HBsAg negative by ARCHITECT HBsAg test.
HBsAg seroconversion rate | 48 weeks
  HBsAg seroconversion rate at 48 weeks off treatment follow-up in patients with HBsAg loss
Surface antibody disappearing rates | 48 weeks
  Surface antibody disappearing rates at 48 Weeks off treatment Follow-up in Patients with HBsAg loss
Viral reactivation rate | 48 weeks
  Viral reactivation rate (HBV DNA > 20 IU/ml) at 48 weeks off treatment in patients with HBsAg loss

CONTACTS AND LOCATIONS:
Locations (1):
- Fahong Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided